CLINICAL TRIAL: NCT02411006
Title: Prediction and Pre-commitment Mailings for Medication Adherence
Brief Title: Effect of Reminders on Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: H14P001
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

ARMS (6):
- Usual care control (No Intervention): No intervention, just usual care from the insurance company
- Reminder control (Experimental): Send a reminder to subjects every month
  Interventions: Behavioral: Reminder
- Anonymous prediction (Experimental): Ask subjects to anonymously predict their upcoming medication adherence
  Interventions: Behavioral: Prediction mailing; Behavioral: Reminder; Behavioral: Anonymity
- Anonymous commitment (Experimental): Ask subjects to anonymously commit to their upcoming medication adherence
  Interventions: Behavioral: Commitment mailing; Behavioral: Reminder; Behavioral: Anonymity
- Identified prediction (Experimental): Ask subjects to predict their upcoming medication adherence and report it
  Interventions: Behavioral: Prediction mailing; Behavioral: Reminder; Behavioral: Identification
- Identified commitment (Experimental): Ask subjects to commit to their upcoming medication adherence and report it
  Interventions: Behavioral: Commitment mailing; Behavioral: Reminder; Behavioral: Identification

INTERVENTIONS:
Behavioral: Prediction mailing — Ask people to predict their upcoming medication adherence
  Arms: Anonymous prediction; Identified prediction
Behavioral: Commitment mailing — Ask people to commit to their upcoming medication adherence
  Arms: Anonymous commitment; Identified commitment
Behavioral: Reminder — Remind people to take their medicine
  Arms: Anonymous commitment; Anonymous prediction; Identified commitment; Identified prediction; Reminder control
Behavioral: Anonymity — Keep patient predictions and commitment anonymous
  Arms: Anonymous commitment; Anonymous prediction
Behavioral: Identification — Ask patients to report their predictions and commitments
  Arms: Identified commitment; Identified prediction

SUMMARY:
The investigators seek to increase medication adherence of subjects. The investigators will send mailings to customers of an insurance company, asking them to predict or commit to a certain level of behavior. The investigators will measure whether this increases medication adherence.

DETAILED DESCRIPTION:
The investigators seek to increase medication adherence of subjects. The investigators will send mailings to customers of an insurance company, asking them to predict or commit to a certain level of behavior. The investigators will measure whether this increases medication adherence. The investigators will send mailings to subjects once per month, and elicit responses via mail, phone, and web surveys.

ELIGIBILITY:
Inclusion Criteria:

* customers of the investigators' insurance company partner

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47088 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Medication refills | 6 months
  frequency of refilling medication

SECONDARY OUTCOMES:
Hemoglobin A1C | 6 months
LDL cholesterol | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Milkman, Ph.D, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Dai H, Mao D, Volpp KG, Pearce HE, Relish MJ, Lawnicki VF, Milkman KL. The effect of interactive reminders on medication adherence: A randomized trial. Prev Med. 2017 Oct;103:98-102. doi: 10.1016/j.ypmed.2017.07.019. Epub 2017 Jul 24. PMID 28751176